CLINICAL TRIAL: NCT00854750
Title: Modeling and Treating the Pathophysiology of Demyelination in Multiple Sclerosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor Enrollment- schedule of assessments too complex and time-consuming.
Sponsor: Elliot Frohman (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Elliot Frohman, Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACTHAR version 1.0
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis, hx of unilateral ON, evidence of thermal sensitivity, and no evidence of an ocular motor syndrome; Multiple Sclerosis, no evidence of ON, and evidence of thermal sensitivity; Healthy age/gender matched controls
MeSH Terms: conditions — Multiple Sclerosis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ACTHAR- placebo first (Experimental): Placebo, 20 mg, 40 mg, 80 mg
  Interventions: Drug: ACTHAR
- ACTHAR- placebo second (Experimental): 20mg, Placebo, 40 mg, 80mg
  Interventions: Drug: ACTHAR
- ACTHAR- placebo third (Experimental): 20 mg, 40 mg, Placebo, 80 mg
  Interventions: Drug: ACTHAR
- ACTHAR- placebo fourth (Experimental): 20 mg, 40 mg, 80 mg, Placebo
  Interventions: Drug: ACTHAR

INTERVENTIONS:
Drug: ACTHAR — SQ weekly injections
  Arms: ACTHAR- placebo first
Drug: ACTHAR — SQ weekly injections
  Arms: ACTHAR- placebo second
Drug: ACTHAR — SQ weekly injections
  Arms: ACTHAR- placebo third
Drug: ACTHAR — SQ weekly injection
  Arms: ACTHAR- placebo fourth

SUMMARY:
The investigators principal hypothesis is that INO and optic neuritis are objective, quantitative, and reproducible models for corroborating the hypothesis that changes in core body temperature are associated with the reversible and stereotypic decay in axonal conduction and that ACTHAR can serve to prevent such changes. The application of ocular motor and optic nerve measures appears to constitute a useful paradigm to detect and monitor responses to therapeutic strategies that stabilize nerve cell membranes in response to temperature induced decay in axonal conduction mechanisms, with implications on activities of daily life that are dependent upon vision (reading, driving, walking, work performance).

DETAILED DESCRIPTION:
A quantum leap forward in our understanding of MS pathophysiology was provided by the discovery of myelin by Louis Ranvier in 1878, and by Pierre Marie who first suggested in 1892 that demyelination represented a critical element in MS pathology.1 In 1925 Lord Edgar Douglas Adrian reported the first electrical recordings of nerve transmission.2 Ultimately six Nobel prizes were awarded for contributions directly related to the characterization of the nerve impulse and the role played by myelin, a monumental achievement of modern biology.

While working at the University of Otago in New Zealand, Dr. W. Ian McDonald (who passed away on December 13, 2006) was the first to provide objective evidence that demyelination in MS was associated with a corresponding change in the transmission of electrically coded messages within nerve axons.3-5 He noted that the disruption of myelin led to a reduction in axonal cross sectional area and thereby a reduction in conduction velocity, loss of saltatory conduction, with a predilection to conduction block. Understanding this conspicuous aspect of MS pathophysiology allows us to predict many of the reversible symptoms described by our patients, particularly those that are provoked or intensified by elevated ambient or core body temperature, exercise, and infection. Such processes appear to compromise the safety threshold for high fidelity nerve transmissions. This phenomenon was also recognized clinically by Wilhelm Uhthoff in 1899, when he evaluated optic neuritis patients who experienced reversible and stereotypic alterations in vision after exercise or exposure to heat.6 MS exacerbations (via inflammation, edema, and demyelination) and sustained progression of disability (via gliosis, sustained demyelination, and neurodegeneration) represent formidable challenges of the disease process that have partially yielded to a series of disease modifying therapeutic strategies.7 However, in most patients, bona fide exacerbations typically occur infrequently (perhaps a few per year, even in those not using treatment), and disability progression takes time (many years in most). Alternately, fluctuations in neuronal activity can be induced by a variety of factors with great frequency and variability (provoked over minutes, hours, days, or weeks) and correspondingly results in a compromise of functional capabilities such as vision, reading, driving, walking, work performance, cognitive processing, and the execution of activities of daily living. In essence, these frequent, transient, typically stereotypic and reversible physiologic changes constitute a major component of MS related disability.

Notwithstanding the important achievement of validating the favorable effects of disease modifying agents in MS, a major and recalcitrant challenge, that should be at the forefront in MS therapeutics, is a focus on reducing the consequences of symptoms collateral to the disease process. Such symptoms include fatigue, weakness, gait dysfunction, spasticity, heat intolerance, pain, cognitive changes, sensory disturbances, bowel, bladder, sexual dysfunction, depression, and hopelessness.8 While the underpinnings of these complaints are manifold, changes in axonal conduction mechanisms now represent a well-recognized and cardinal feature of MS pathophysiology.

A deeper understanding on how novel interventions might serve to enhance the axonal 'safety factor' to thermal perturbations (ambient, surface, and core body temperature) could lead to the identification of new treatment strategies for enhancing physiologic performance in CNS pathways involved in the organization of physical and intellectual capabilities. An important randomized controlled study systematically demonstrated the long-term benefits of acute and chronic cooling on objective as well as patient reported measures of neurologic function.9 It would be important to also understand how active heating impacts upon similar measures, and whether preemptive cooling is protective in response to a heat stress.

We propose that neuro-ophthalmologic hallmarks of MS, INO (an ocular motor syndrome) and optic neuritis (a visual sensory syndrome), can be studied with objective methods (infrared oculography and VEPs respectively) to better understand the factors that provoke or prevent the reversible conduction changes in demyelinated axons, within highly discrete tract systems and whether a specific drug treatment, ACTHAR Gel, can mitigate heat induced worsening of ocular motor and anterior visual system dysfunction. Such studies would appear to be germane to the development of new treatment approaches focused on optimizing the fidelity of axonal conduction in demyelinated pathways, and providing elusive outcome measures for some Phase II trials. Education efforts to inform patients and health care providers on the pervasive nature of thermally induced symptoms in MS (and the potential impact on daily activities), could lead to effective strategies to enhance performance and safety. There has been a paucity of research and education on this very conspicuous and important aspect of MS and its impact upon patients, families, and the workplace.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has clinically or laboratory supported Multiple Sclerosis with evidence of INO by quantitative neurophysiologic criteria or has a history of ON.
2. Subject is between the ages of 18-65.
3. Subject is able to understand the demands of the protocol, has had any questions answered and has voluntarily signed the informed consent prior to any study procedures.
4. Subject has a peak saccadic acceleration ratio (abducting eye/adducting eye) of greater than 2S.D. above the mean derived form a normal control group.
5. Subject is otherwise in good health, based on complete medical history and physical examination, including vital signs and ECG.

Exclusion Criteria:

1. Subject is a pregnant female (as determined by a urine pregnancy test), a lactating female, or a female of child-bearing potential, not sterilized and not using one of the following methods of birth control: oral or injectable contraceptive agent, implantable contraceptive device, or barrier method.
2. Subject has a history of hypertension or diabetes.
3. Subject has known allergy to ACTH.
4. The subject has any medical condition, including psychiatric disease that might interfere with the interpretation of the results or with the conduct of the study.
5. Subject has a history of drug or ethanol abuse within the past year.
6. Subject has a history of ischemic heart disease.
7. Subject has received an investigational drug within 30 days of screening.
8. In opinion of investigator, subject is unlikely to complete study for any reason.
9. The subject has abnormal clinical laboratory values or an abnormal ECG, without approval of the study monitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To determine if preemptive cooling provides protection against worsening of INO and its effect on reading, with body heating. | 8-10 weeks for each patient

SECONDARY OUTCOMES:
To determine whether changes in core body temperature has an impact on patient reported measures of vision (high and low contrast acuity) and reading acuity and speed. | 8-10 weeks per patient

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Frohman, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States